CLINICAL TRIAL: NCT01294982
Title: Phase II, Randomized, Double-blind, Placebo-controlled Trial of the AOBO-001 for the Treatment of Overactive Bladder With Symptoms of Urge Urinary Incontinence and Frequency
Brief Title: Study of AOBO-001 for Overactive Bladder With Urge Urinary Incontinence and Frequency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Oriental Bioengineering, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20100011031
Record Dates: First submitted 2011-01-04; First posted 2011-02-14 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Overactive Bladder
Keywords: OAB; Over Active Bladder; overactive bladder; Urinary Urge Incontinence; Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1.6 g AOBO-001 Group (Experimental): AOBO-001 400 mg Oral Capsules
  Interventions: Drug: AOBO-001
- 3.2 g AOBO-001 Group (Experimental): AOBO-001 400 mg Oral Capsules
  Interventions: Drug: AOBO-001
- Placebo (Placebo Comparator): Matching Placebo Capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AOBO-001 — AOBO-001 400 mg Oral Capsules (1.6 g dose) twice daily
  Arms: 1.6 g AOBO-001 Group
Drug: AOBO-001 — AOBO-001 400 mg Oral Capsules (3.2 g dose) twice daily
  Arms: 3.2 g AOBO-001 Group
Drug: Placebo — Placebo Oral Capsules twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and effectiveness of the study product, AOBO-001, when taken by adults with symptoms of overactive bladder. AOBO-001, is experimental, which means that the U. S. Food and Drug Administration (FDA) has not yet approved it for use. AOBO-001 has been approved in China as a prescription drug product to treat bedwetting in children. AOBO-001 is also approved in Hong Kong as a dietary supplement to improve quality of life for people with urinary incontinence. AOBO-001 is a botanical (from a plant) product. It is prepared from the seeds of Xanthoceras sorbifolia bunge plant, which is a flowering tree grown in Northern China. Approximately 60 subjects who are 18 years of age and older are expected to participate in this study at up to 8 investigational sites. Each subject will complete 6 visits to the study site over a 14-week period. Subjects will consume 8 capsules of the assigned test product twice daily (that is, 16 capsules daily). Capsules will be taken with at least 6 ounces of water approximately 30 minutes before breakfast and 30 minutes before dinner. If a subject qualifies, he/she will be randomly (by chance) assigned to one of three study treatment groups. Subjects in one group will consume capsules containing a daily dose of 3.2 grams of AOBO-001; a second group will consume capsules containing a daily dose of 6.4 grams of AOBO-001; and a third group will consume capsules containing a placebo (no active ingredients). Subjects will have a 2 in 3 chance of being assigned to an active study treatment group. Neither the subject nor the study doctor will know to which study treatment group the subject has been assigned, but this information is available in case of a medical emergency. There will be a time during the study dosing schedule when all subjects will consume capsules containing a placebo (no active ingredients). Subjects will not be told when they are receiving the placebo.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled Phase 2 clinical trial will evaluate the safety and efficacy of AOBO-001 in adults with overactive bladder. The primary objective of this study is to evaluate the efficacy of AOBO 001 compared with placebo on the basis of the change from baseline in average number of micturition episodes per 24 hours from the 3-day diaries and average number of urge urinary incontinence episodes per 24 hours from the 3 day diaries during the double-blind treatment period in adult patients with OAB. Secondary efficacy objectives are to evaluate the efficacy of AOBO-001 compared with placebo on the basis of the number and severity of urgency episodes by using the Patient's Perception of Intensity of Urgency Scale (PPIUS), nocturia episodes, volume voided per micturition, and Patient Perception of Bladder Condition (PPBC) global assessment measure. An additional secondary objective is to evaluate the safety and tolerability of AOBO-001 compared with placebo.

Eligible patients will be randomized in equal proportions to double-blind treatment with AOBO 001 1.6 g twice daily (3.2 g daily), AOBO-001 3.2 g twice daily (6.4 g daily) or placebo capsules twice daily.

Efficacy assessments include urinary diary assessments, including the number of micturitions (daytime, nighttime), number of urge incontinence episodes, number/grading of urgency episodes (Patient's Perception of Intensity of Urgency Scale or PPIUS), and volume of voided urine; and Patient Perception of Bladder Condition (PPBC) questionnaire. Safety assessments include post-void residual urine volume measured by bladder scan; vital signs, 12-lead ECGs, complete or brief physical examinations, clinical laboratory safety tests, and treatment-emergent adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female aged 18 years or older and provides written informed consent;
2. Patient has had symptoms of OAB, including urinary frequency, urgency or urge incontinence, for at least 3 months prior to the screening visit;
3. Patient is compliant with completing 3 consecutive days of the urinary diary each week and at least 85% compliant with taking placebo capsules during the 2-week placebo run-in period;
4. Patient experiences an average micturition frequency of ≥8 times per a 24-hour period based on the 24-hour average of 3 consecutive days of urinary diary data during the last week of the 2-week placebo run-in period;
5. Patient has had at least 4 episodes of incontinence over a 3 consecutive day urinary diary period during the 2-week placebo run-in period; and
6. Patient has had at least 4 episodes of urgency (PPIUS Grade 3 or 4) with or without incontinence over a 3 consecutive day urinary diary period during the 2-week placebo run-in period.

Exclusion Criteria:

1. Patients with known allergy to plants of Sapindaceae family, including maple syrup, litchi (Litchi chinensis), rambutan (Nephelium lappaceum), longan (Euphoria longana), ackee (Blighia sapida) and Spanish Lemon (Melicoccus bijugus).
2. Pregnant women or women who intend to become pregnant during the study or women of childbearing potential who are sexually active and practicing an unreliable method of birth control or will be lactating during the study. Reliable contraceptive methods are intra-uterine devices, double-barrier method (condom with spermicide), contraceptive pills of combination type, hormonal implants and injectable or patch contraceptives;
3. Clinically significant outflow obstruction (at the discretion of the investigator);
4. Significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor, as determined by the investigator;
5. Patient with indwelling catheters or practicing intermittent self-catheterization;
6. Evidence of a symptomatic urinary tract infection, chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs;
7. Non-drug OAB treatment such as bladder-training, biofeedback and pelvic floor exercises are permissible if established at least 4 weeks prior to study start and intended to be continued throughout the study; electrostimulation therapy is not permissible at any time;
8. Use of drugs intended to treat urinary incontinence, such as darifenacin (Enablex), fesoterodine (Toviaz), oxybutynin (Ditropan, Ditropan XL, Oxytrol), solifenacin (Vesicare), tolterodine (Detrol, Detrol LA), and trospium (Sanctura, Sanctura XR);
9. Any clinically significant condition, which in the opinion of the investigator makes the patient unsuitable for the trial, including without limitation, major cardiovascular or cerebrovascular event (e.g., myocardial infarction, stroke, unstable angina, transient ischemic attacks) within the past year, major neurological disorders (e.g., paralysis or neuropathies, multiple sclerosis), major psychiatric diseases (e.g., major depression, generalized anxiety, psychosis), unstable or poorly controlled chronic diseases (e.g., uncontrolled moderate to severe hypertension or poorly controlled diabetes mellitus), and moderate to severe renal or hepatic disease;
10. Participation in any clinical trial within 30 days prior to randomization;
11. Women who suffer from undiagnosed vaginal bleeding;
12. Employees of AOBO, third parties associated with the study, or the study site; and
13. Patient who did not complete the urinary diary (3 consecutive days of valid urinary diary data each week) and did not take placebo run-in study medication (at least 85% compliance) according to the instructions during the placebo run-in period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in average number of micturitions per 24 hours from 3-day urinary diaries compared to baseline | Endpoint (up to 12 weeks of double-blind treatment)
  Change in the average number of micturitions per 24 hours from the 3-day diaries from baseline to endpoint of the 12 week double-blind treatment period.
Change in average number of urge incontinence episodes per 24 hours from 3-day urinary diaries compared to baseline | Endpoint (up to 12 weeks of double-blind treatment)
  Change in average number of urge urinary incontinence episodes per 24 hours from the 3-day diaries from baseline to endpoint of the 12 week double-blind treatment period.

SECONDARY OUTCOMES:
Change in volume voided per micturition compared to baseline | Endpoint (up to 12 weeks of double-blind treatment)
  Volume voided per micturition over 24 hours.
Change in intensity of urgency episodes compared to baseline | Endpoint (up to 12 weeks of double-blind treatment)
  Intensity of urgency episodes, PPIUS grade 3+4, intensity of urgency episodes, PPIUS grades 0-4, and maximum urgency intensity at void episodes (PPIUS grades 0-4) per 24 hours.
Change in daytime and sleeptime micturitions compared to baseline | Endpoint (up to 12 weeks of double-blind treatment)
  Number of daytime and sleeptime (nocturia) micturition episodes per 24 hours.
Change in weekly urge incontinence episodes compared to baseline | Endpoint (up to 12 weeks of double-blind treatment)
  Number of urge urinary incontinence episodes per week.
Change in PPBC score compared to baseline | Endpoint (up to 12 weeks of double-blind treatment)
  Patient Perception of Bladder Condition (PPBC) score.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | During double-blind treatment phase
  Treatment-emergent adverse events including subject reporting, clinical observations, and clinically significant abnormal findings as measured by bladder scan, vital signs, 12-lead ECGs, complete or brief physical examinations and clinical laboratory safety tests.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Du, MD, PhD, Study Director — American Oriental Bioengineering, Inc.
Locations (5):
- United States (5):
  - Coastal Clinical Research, Mobile, Alabama
  - Palm Beach Research Center, West Palm Beach, Florida
  - Heartland Research Associate, LLC, Newton, Kansas
  - Myron I. Murdock M.D. LLC, Greenbelt, Maryland
  - Regional Clinical Research, Inc, Endwell, New York